CLINICAL TRIAL: NCT05151094
Title: Registry of Hospitalized Patients in University Hospital Dubrava Respiratory Center
Acronym: COVID-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Marko Lucijanić, Study Director, University Hospital Dubrava
Other Study IDs: 2021/2503-04
Record Dates: First submitted 2021-09-20; First posted 2021-12-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Covid19; Thrombosis; Bleeding; Sepsis; Mechanical Ventilation Complication; Inflammatory Response
MeSH Terms: conditions — COVID-19; Thrombosis; Hemorrhage; Sepsis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Remdesivir exposure: Patients treated with remdesivir due to the COVID-19 infection
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation of clinical outcomes and comparison to non-treated patients

SUMMARY:
Aim of this project is to understand clinical features, clinical outcomes and efficacy and safety profiles of different therapies by analyzing a cohort of COVID-19 patients hospitalized and treated in a tertiary-level institution, University hospital Dubrava. Patients' clinical and laboratory characteristics, drug exposure and outcomes are obtained by analysis of written and electronical medical records.

DETAILED DESCRIPTION:
University Hospital Dubrava has been completely repurposed during the COVID-19 pandemic to become high volume COVID-19 tertiary institution. Establishment of hospital registry project is necessary to properly understand disease characteristic, related outcomes and real-life treatment patterns. Registry provides a fundamental framework for future upgrading with emerging or retrogradely obtained specific data that will substantially facilitate understanding of COVID-19 in the context of other specific diseases, therapies and procedures. Large comprehensive database will provide sufficient statistical power to allow for investigation of large number of subgroups and existence of interactions between different variables. Assessment of large number of clinically important outcomes (mortality, occurrence of venous and arterial thromboses, major bleeding, bacteriemia, incidence of mechanical ventilation and intensive care unit admission) is necessary to put any investigated parameter in the proper efficacy and safety context.

ELIGIBILITY:
Inclusion Criteria:

* all hospitalized patients positive for COVID-19

Exclusion Criteria:

* none

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients that were hospitalized in our institution due to the COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | At 30-days from hospital admission
  Incidence of death from any cause

SECONDARY OUTCOMES:
Incidence of venous or arterial thrombotic events | At 30-days from hospital admission
  Incidence of arterial or venous thromboses proven by objective imaging (ultrasound, computerized tomography, magnetic resonance imaging, scintigraphy) and laboratory (troponin) methods.
Incidence of major bleeding | At 30-days from hospital admission
  Incidence of bleeding events that can be classified by the International Society on Thrombosis and Haemostasis criteria as major bleeding.
Incidence of bacteriemia | At 30-days from hospital admission
  Incidence of positive blood cultures that were taken based on clinical suspicion for bacterial co-infection.
Incidence of mechanical ventilation | At 30-days from hospital admission
  Incidence of mechanical ventilation use required for deteriorating respiratory function.
Incidence of intensive care unit admission | At 30-days from hospital admission
  Incidence of intensive care unit admission required for intensive/critical level of care.

CONTACTS AND LOCATIONS:
Overall Officials: Marko Lucijanic, MD PhD, Study Director — University Hospital Dubrava
Locations (1):
- University Hospital Dubrava, Zagreb, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No